CLINICAL TRIAL: NCT02493842
Title: Natural Sensory Feedback for Phantom Limb Modulation and Therapy
Brief Title: Direct Nerve Stimulation for Treatment of Phantom Limb Pain
Acronym: EPIONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other); University of Lausanne Hospitals (Other); University of Freiburg (Other); Université Montpellier (Other); Lund University (Other); Indiana University School of Medicine (Other); Novosense AB (Industry); Mxm-Obelia (Industry); Ecole Polytechnique Fédérale de Lausanne (Other); Universitat Autonoma de Barcelona (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIONE-602547-5; no. 602547 (Other Grant/Funding Number: FP7-HEALTH-2013-INNOVATION)
Record Dates: First submitted 2015-06-22; First posted 2015-07-10 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Phantom Limb Pain
Keywords: Nerve Stimulation; Neuroplasticity; Sensory Feedback
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Invasive nerve stimulation (Experimental): Invasive nerve stimulation using the following experimental devices
  1. Transverse Intrafascicular Multichannel Electrode for human (TIME-4H)
  2. The STIMEP stimulator
  3. The EPIONE Psychophysical Testing Platform software for stimulator control
  Nerve stimulation therapy is provided while providing visual guidance to the subject and without the use of hand prosthetic devices
  Interventions: Device: Transverse Intrafasicular Multichannel electrode (TIME)

INTERVENTIONS:
Device: Transverse Intrafasicular Multichannel electrode (TIME) — Peripheral nerve stimulation is conducted with Transverse Intrafasicular Multichannel electrode (TIME) version 4 electrodes to induce sensory sensations from the phantom hand, while subject is virtualizing a movement or event which may cause the specific sensation.

SUMMARY:
Background:

Phantom limb pain (PLP) develops in 50-80% of subjects who have a limb amputated. It is not well known what causes PLP to develop and the current treatments have been shown to be largely ineffective. Resent research, however, have indicated that cortical reorganizing occurring after amputation of the cortex areas related to the missing limb may be related to the development of PLP. Furthermore, the research indicated that by providing meaningful sensory input coming from the phantom limb the PLP may be alleviated and the cortical organization normalized.

Aim:

The CIP described in the current application, is part of a the EU-project "EPIONE", which aims to investigate if and how cortical normalization and PLP alleviation can be induced by providing phantom limb sensations (sensations which seems to originate from the missing limb) in hand amputated subjects.

Method:

In the current study, which will take place at Aalborg University Hospital (AUH), 2-4 hand amputated subjects experiencing severe PLP will implanted with interneural nerve electrodes in the arm stump for up to one year.

Therapy will be evaluated in two stages, first during a standardized four week phase where the subject receives daily therapy. If the therapy is shown to be effective, therapy may be reinitiated during a second longer therapy phase.

During the therapy sessions, selective nerve stimulation will be performed. The amputee will experience this as sensations (movement, touch, temperature, vibration etc.) originating from the phantom limb. While implanted, we will investigate how well we can induce these sensations and we will provide a stimulation therapy, which consist of stimulation activities which requires the subject to focus on the evoked sensations. Prior to, during a and following therapy a series of assessments (standardized across all EPIONE partners to enable comparison) will be conducted to relate therapy with PLP, cortical organization, the mental state etc. of the subject.

Expected outcome:

The stimulation therapy is expected to alleviate PLP and induce cortical normalization. The experience we gain might be used for deriving clinical guidelines on how to treat PLP.

DETAILED DESCRIPTION:
The study will be carried out in two parts. The first part will function as a pilot part where the investigators will seek to get experience with, e.g., stimulation procedures: Which therapies activities and stimulation parameters do the participants feel are the most intuitive (i.e., most effective reintroducing the phantom hand into the body image of the amputee) and thus might be expected to be most effective in normalizing the cortical organization and alleviating PLP.

After part 1 the data will be analyzed together with the international partners (no participants identifiable data will be shared) and the shared experiences will be used to adjust the activities of part two.

The experiment is conducted in the following phases:

1. Startup
2. Pre-screening
3. Baseline and entry
4. Implantation (defined as week 0)
5. Therapy
6. Outcome
7. Follow-up
8. Repetition. Redo phase 3 to 7 with longer therapy phase durations only

Procedures during phases 1 to 7 (weeks -5 to 12) are standardized across international EPIONE partners (which carry out different interventions, but similar assessments), to enable comparison between treatment modalities. At AUH, if therapy is shown to be effective during phase 1-7, the investigators will repeat the initial phases 3 to 7, but with a longer therapy phase, to investigate the effect of long term stimulation therapy. TIME-4H electrodes will not be left implanted for a longer duration than one year.

During the different phases of the study a collection of assessment methods is conducted to monitor the effect of stimulation therapy on the amputee's level of perceived PLP and cortical organization. In addition, the psychological state of the subject, the strength and type of the non-painful phantom limb sensations are also assessed to provide a more detailed view on the possible effects of the stimulation therapy.

The experiment will be conducted as a series of case studies where the effect of the stimulation therapy in a participant is compared with the PLP sensations the same subjects perceived before initiating the therapy. Therefore, only amputees who are in a stable state (e.g., not newly amputated subjects) are included in the study.

No placebo or blinding is performed as the participant can feel the stimulation and also has to be mentally active involved in performing "phantom limb movements" when receiving stimulation therapy.

Phases 1-7 for each subject (week -3 to week 12, week = 0 is implantation) are performed according to the experiment protocol defined in collaboration with international partners. Phase 8, has been defined by AUH, and is constituted by a repetition of the phases 3-7, where the treatment phase has been prolonged.

Phase 1: Startup The participant is invited to a meeting with the principal investigator and one of the senior researchers involved in the study to be informed about the experiment. Only the PI, who is a medical doctor, will be allowed to answer health and medical related questions.

Phase 2: Pre-screening This phase is conducted before the start of the experiment but after the subject has signed the informed consent form and the authority form, the latter granting representatives from Danish Health and Medicines Agency access to the study data and patient record for control purposes. Via questionnaires, tests and interviews it is evaluated if the participant fulfills the inclusion criteria in relation to physical health (able to undergo surgery), depression, normal range of IQ and PLP. The principal investigator will evaluate the results and decide whether the participant should be included or excluded.

Phase: Baseline and entry The baseline and entry phase aims to determine the stability and intra-subject variability of the pain sensations without treatment. The measure control for the daily variability in pain, assessment scoring variability, site-to-site variability and inter subject variability in the "before intervention" state. These variances will be used in the analysis to estimate baseline noise in the measure.

A second rationale for the repetition of these measures in this phase is to trap any effect that might come out of running the assessment, e.g., due to the increased attention on PLP.

If the participants live close to AUH, these assessments will be conducted at AUH under supervision of experimenters. If it is unpractical for the participants to attend the daily sessions at AUH, the subject may conduct them at home after receiving adequate training and while being in regular contact with an experimenter. If performed at home, assessments (questionnaire) may be filled out by the subjects on printed-out versions or using a laptop with the Psychophysical Testing Platform installed using a participants specific login with accompanying functional restrictions.

In addition to the questionnaire used for quantifying the perceived phantom limb pain and sensation, the last week before implantation includes the application of cortical mapping methods (EEG, SEP and fMRI).

During all phases of the study the subject is required to fill out a diary before going to bed about the development of PLP during the day.

Phase 3: Implantation Surgical implantation of the TIME-4H electrodes is conducted under full anesthesia. During the operation, the median and the ulnar nerves are freed through an incision of 20 cm on the medial aspect of the upper-arm. The fascicles of both nerves are dissected free for a couple of centimeters at the level where the TIME-4H electrodes are to be implanted. Four TIME-4H electrodes are pulled in to the fascicles of the nerves using the attached needle and thread, two TIME-4H in each nerve. The electrode are anchored to the nerve using the dedicated anchoring points of the TIME-4H (seen on figure 4 (B)). After placing the electrodes the electrical integrity of each TIME-4H electrode is tested, before closing the wound. Lead out wires are lead out through the skin and the wound is closed. During surgery the participant is treated with prophylactic antibiotics. Prophylactic antibiotics are not administered later in the study due to the risk of the development of resistance.

After the implantation the subject is offered to stay at Patienthotellet to enable routine assessment of the surgical outcome as long as the PI judges it necessary.

Wound treatment While the electrodes are implanted, the subject will routinely have the wound where the wires exit the arm cleaned and treated to reduce the risk of infection. This will be conducted by a nurse who is member of the project group.

The participant will receive training in treating/cleaning the wound and also in what symptoms to be aware of. During phases of the study where the subject does not attend daily therapy sessions and thus is not in daily face-to-face contact with the project team, the participant may for shorter periods perform the wound treatment him/herself.

Phase 5: Therapy Phantom limb pain and sensations are assessed via questionnaire prior to and following the stimulation therapy. Several assessments are conducted during this phase with the purpose of characterizing the sensations which can be evoked and to provide sensory stimulation therapy with the aim of alleviating the phantom limb pain.

* PsyP-Map (B): Stimulation is conducted using each of the individual contact sites and different combinations of the implanted TIME-4H with the purpose (1) of determining suitable (above sensation threshold and below pain threshold) stimulation parameters (intensity, pulse width etc.) and (2) of mapping the perceived location and type of the sensations evoked.

  o Will be conducted once every week; each session will last approx. 2 hours.
* Stimulation therapy: Stimulation is performed with the aim of inducing meaningful sensory input to the subject and thereby inducing a normalization of the cortical organization and alleviation of PLP. This is sought accomplished by performing activities which reintroduce the missing limb into the subject's body image:

  * The subject is instructed to imagine performing a movement or sensation indicated on the subject computer screen with the phantom hand. During this "movement" the experimenter will seek to evoke relevant sensations via electrical stimulation.
  * The therapy session will be conducted once every weekday; each session will last approx. 2 hours.

If the results indicate that the therapy was effective and the subject is interested in continuing the therapy, the TIME-4H electrodes are left implanted during the outcome and follow-up phase. However, no stimulation therapy is performed during these phases.

An fMRI examination is scheduled to be carried out at the end of the therapy phase. The TIME-4H is currently being tested for MR compatibility, and the result is expected in March 2015. If the TIME-4H is compatible, the fMRI examination will be conducted as planned. If it is not compatible, the fMRI examination will be conducted when the TIME-4H has been explanted.

Phase 6: Outcome After four weeks of therapy a series of assessments are performed to assess the effect of therapy.

No stimulation therapy is conducted during the outcome and the following follow-up phase.

Phase 7: Follow-up During the follow-up phase it is assessed how long time it takes for any effects pain alleviating effect of the therapy to wear off.

The frequency of the follow-up assessment will be dependent on whether the therapy is effective in the individual subjects (entry assessments compared with outcome assessments). If effective, follow-up assessments are conducted one time each week, 2, 4 and 8 weeks after ended therapy. If deemed ineffective, follow-up assessments are only conducted 4 weeks after ended therapy (week 8).

At the end of the follow-up phase the procedures standardized between the EPIONE international partners end, and partners decide individually how to proceed.

Phase 8: Repetition of therapy At AUH, in the case that the applied stimulation therapy reduces the PLP of the subject and the subject is interested in continuing the therapy, the therapy may be reinitiated by repeating the procedures of phase 3 to7, however, with a longer therapy period.

The study duration for a subject will be limited by the maximum TIME-4H implantation duration, which has been set to one year maximum, and later in the study the overall termination of experimental activities in the EPIONE study.

Recognizing the potential long duration of the study and the large effect daily therapy sessions will have on the subject's everyday life, especially for subjects living far from AUH, the therapy will be adjusted in terms of frequency (e.g., one time weekly) and duration (hours per session) to suit the subject, while aiming at the administration of enough therapy to induce a sufficient PLP alleviating effect.

Explantation In the event of infection, blushing, swelling, pain or other complications which render continuous implantation impossible, the electrodes will be explanted and the subject treated with antibiotics.

Explantation of the TIME-4H electrodes may be conducted at the end of the therapy phase if the therapy is unsuccessful or if the subject does not wish to continue.

If the subject wishes to continue the therapy, the maximal allowed implantation time will be 1 year.

Explantation will be carried out under full anesthesia. Access is obtained via an insertion made through the skin on the medial side of the upper arm. The TIME-4H electrodes are dissected free, thread cut and the implant pulled out of the nerve and removed. Following the explantation normal wound treatment will be conducted and the stitches removed according to standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman >18 yrs and < 70 yrs.
* Unilateral transradial amputation.
* Other treatments for PLP tried with poor results
* Patient accepts the study protocol as explained by the physician.
* The subject must experience intractable PLP higher than 6 on a Visual Analog Scale (VAS) from 0-10. The frequency of PLP attacks must present itself more than once a week.
* Amputation should be in the chronic, stable phase, such that the stump has healed and the person apart from experiencing phantom pain is healthy and able to carry out the experiment.

Exclusion Criteria:

* Cognitive impairment
* Current or prior psychological impairments: major personality disturbance (i.e., borderline, antisocial), major depression, bipolar I.
* Pregnant (if fertile woman: assessed via a pregnancy test) or not using contraception accepted by the authorities during the study
* Breastfeeding women cannot participate in the study
* History of or active substance abuse disorder.
* Acquired brain injury with residual impairment
* Intellectual Disability (IQ < 70)
* Current or prior neurological or musculoskeletal disease
* Current or prior dermatological conditions
* Persons with other diseases that may affect the function of the nervous system, e.g., diabetes, HIV or renal failure.
* Subjects who will not be able to have an fMRI examination conducted because of metal implants such as: pacemakers, artificial joints, bone screws.
* Subjects who suffer from claustrophobia and who are unable of having an fMRI examination conducted (the examination requires the subject to lie inside a narrow space in the MRI machine).
* Subjects cannot participate in other clinical studies and/or tests of medical devices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Phantom limb pain | Change in pain perception over 3 -15 months. (Time frame is dependent on effect of treatment)
  The pain intensity will be assessed using a visual analog scale (VAS) analog scale (VAS), the neuropatic pain sympton inventory (NPSI), the brief pain inventory interference scale (BPSI)
Cortical reorganization | Change in pain perception over 3 -15 months. (Time frame is dependent on effect of treatment)
  The cortical response to peripheral stimulation will be tracked using MRI MRI and EEG.

SECONDARY OUTCOMES:
Cortical reorganization | Change in pain perception over 3 -15 months. (Time frame is dependent on effect of treatment)
  The cortical response to peripheral stimulation will be tracked using EEG
Phantom limb pain | Change in pain perception over 3 -15 months. (Time frame is dependent on effect of treatment)
  The pain symptoms wil be assessed using the neuropatic pain symptom inventory (NPSI)

CONTACTS AND LOCATIONS:
Overall Officials: Preben Sørensen, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark